CLINICAL TRIAL: NCT02667756
Title: Identification of Prognostic Biomarkers for Osteoarthritis Risk Following Knee Injury: the Knee Injury Cohort @ the Kennedy Study
Brief Title: Predicting Osteoarthritis Risk Following Knee Injury.
Acronym: KICK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Fortius Clinic (Other); BUPA Cromwell Hospital, London, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: cro1532; 10/H0805/39 (Other: NRES)
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis; Injury
Keywords: biomarker; inflammation; prognosis; knee
MeSH Terms: conditions — Osteoarthritis; Wounds and Injuries; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples include blood (plasma, serum, whole blood RNA, and where consent given, DNA), urine and where undergoing a relevant clinical procedure to allow sampling, synovial fluid.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-interventional

SUMMARY:
This observational study seeks to identify and validate novel soluble biomarkers (within blood, synovial fluid, urine) which contribute to the prognostic assessment of an individual with an acute knee injury, a group of individuals in which ~50% will progress to symptomatic radiographic knee osteoarthritis (OA).

150 individuals will be followed over 5 years with clinical assessment including validated questionnaires, biological sampling and radiological imaging (X ray, magnetic resonance imaging (MRI)).

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant acute knee injury within 8 weeks of recruitment
* Aged 16-50
* Knee effusion, evident clinically or by MRI
* Evidence on MRI of structural injury (from list of relevant injuries)
* Informed written consent

Exclusion Criteria:

* Knee injured more than 8 weeks prior to recruitment
* Pre-existing advanced radiographic OA (Kellgren Lawrence (KL) grade 3-4) of same side knee at baseline
* Known history of inflammatory/septic arthritis of same side knee
* Knee replacement - previous or planned within 2 years of study start
* Active other (treated) inflammatory disease or infection
* Positive pregnancy test
* Not consenting, or contraindication to provide blood samples:

  * Bilateral mastectomy
  * Bilateral fistulae for renal dialysis
* Unable to give informed written consent in English

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a non-intervention cohort study of subjects who have recently sustained a structural knee injury. Individuals are identified from the practice of a collaborating surgeon (AW) at a number of London sites, several of which are within private practice. Because of the practice of the surgeon investigator, a large number will be sporting professionals, or playing amateur sport at a high level.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-06; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS)-4 score at 2 years | 2 years
  Summary score for KOOS questionnaire

SECONDARY OUTCOMES:
Change from baseline in Kellgren Lawrence grade at 2 years | 2 years
  measured on X ray both knees
Change from baseline in Whole Organ MRI Score (WORMS) at 2 years | 2 years
  measured on MRI both knees
Change from baseline in physical activity level (International Physical Activity Questionnaire, IPAQ) at 2 years | 2 years
  validated activity questionnaire
Change from baseline in KOOS-4 score at 3 months | 3 months
  Summary score for KOOS questionnaire
Change from baseline in KOOS-4 score at 5 years | 5 years
  Summary score for KOOS questionnaire
Change from baseline in Kellgren Lawrence grade at 5 years | 5 years
  measured on X ray both knees
Change from baseline in MRI WORMS score at 5 years | 5 years
  Measured on MRI both knees

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Watt, MD, PhD, Principal Investigator — University of Oxford
Locations (1):
- Kennedy Institute of Rheumatology, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garriga C, Goff M, Paterson E, Hrusecka R, Hamid B, Alderson J, Leyland K, Honeyfield L, Greenshields L, Satchithananda K, Lim A, Arden NK, Judge A, Williams A, Vincent TL, Watt FE. Clinical and molecular associations with outcomes at 2 years after acute knee injury: a longitudinal study in the Knee Injury Cohort at the Kennedy (KICK). Lancet Rheumatol. 2021 Jun 24;3(9):e648-e658. doi: 10.1016/S2665-9913(21)00116-8. eCollection 2021 Sep. PMID 34476411
- See also: Kennedy OA Centre homepage — http://oacentre.kennedy.ox.ac.uk/